CLINICAL TRIAL: NCT03923816
Title: Implications of Variable Intraoperative Fluid Strategies Upon the Hepatic Outcome in Hepatobiliary Surgery
Brief Title: Implication of Fluid Strategies Upon Hepatic Outcome in Hepatobiliary Surgery
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Safwat, specialist, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: fluids and hepatic outcome
Record Dates: First submitted 2019-04-18; First posted 2019-04-23 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Hepatic Complication
MeSH Terms: interventions — Ringer's Lactate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (R) (Experimental): Restrictive fluid strategy:6 mL/kg/h of Lactated Ringer (LR).
  Interventions: Drug: Conservative fluid strategy: 12 mL/kg/h of Lactated Ringer (LR).&Restrictive fluid strategy:6 mL/kg/h of Lactated Ringer (LR).
- Group (C) (Experimental): Conservative fluid strategy: 12 mL/kg/h of Lactated Ringer (LR).
  Interventions: Drug: Conservative fluid strategy: 12 mL/kg/h of Lactated Ringer (LR).&Restrictive fluid strategy:6 mL/kg/h of Lactated Ringer (LR).

INTERVENTIONS:
Drug: Conservative fluid strategy: 12 mL/kg/h of Lactated Ringer (LR).&Restrictive fluid strategy:6 mL/kg/h of Lactated Ringer (LR). — comparison of two intraoperative fluid strategies upon hepatic outcome in hepatobiliary surgery

SUMMARY:
compare the effect of two different protocol of fluid therapy in patients undergoing elective hepatobiliary surgery under general anesthesia regarding hemodynamics and SGPT change pre- and postoperative.

DETAILED DESCRIPTION:
Fluid administration during and after surgery is an essential part of postoperative care to maintain the patients' fluid and biochemical balance. Abdominal surgical procedures are associated with dehydration from preoperative fasting , bowel preparation, and intra- and postoperative fluid and electrolyte loss(1). So, perioperative fluid management has been a topic of much debate over years and has intensified especially over the past several years. The controversies include the type of fluid, the timing of administration and the volume administrated. Following much discussions and ongoing controversy on colloids versus crystalloids(2-5) and the ideal composition of the various intravenous solutions(6-8),the main focus more recently has been on the volume of fluids.

Fluid therapy strategies have been developed and implemented in clinical practice over several decades. The data suggest that aggressive or liberal intraoperative fluid resuscitation is harmful during open abdominal operation, whereas a restrictive fluid protocol has better outcomes, including fewer postoperative complications and a shorter discharge time. (9-11).

However , a restrictive fluid regimen has several limitations (12). Overly restricted or inadequate fluid administration may lead to insufficient intravascular volume, tissue hypoperfusion, cellular oxygenation impairment and potential organ dysfunction(13), prolonged recovery of bowel function, and impair tissue oxygenation, which might ultimately impair wound healing including healing of anastomosis.(14, 15) Recently, The Pleth variability index (PVI) derived from respiratory variations in peripheral perfusion index (PI) has been suggested to be an effective dynamic indicator of fluid responsiveness. Different from other invasive dynamic indices, PVI provides clinicians with a numerical value obtained noninvasively. (16-18) PVI is calculated as [(PImax - PImin)/PImax] X 100, where PImax and PImin represent the maximal and the minimal value, respectively, of the plethysmographic perfusion index (PI) over one respiratory cycle (16, 19). PI is the ratio between pulsatile and no pulsatile infrared light absorption from the pulse oximeter, and it is physiologically equivalent to the amplitude of the plethysmographic waveform (20). A PVI value of >13% before volume expansion discriminated between fluid responders and non-responders with 81% sensitivity and 100% specificity.

An extremely important feature of fluid therapy is ability to modulate inflammatory response in all its aspects with impact on a rate of neutrophil activation and modulation of cytokine and adhesive molecules expression. Isotonic sodium chloride solution and Ringer's lactate solution were shown to have pro-inflammatory properties while so called low volume therapy. Saline solution seems to be the most pro-inflammatory infusion fluid exerting negative impact on both macro- and microcirculation (21). Infusions of high volume of sodium chloride result in elevated serum chloride levels leading to acid-base imbalance and increase of free hydrogen ions (22).

Some available literature data show potential impact of Ringer's lactate therapy on induction of inflammatory response (23) but other reports do not support such phenomenon (24). Acetates similarly to lactates act as buffers and are easily broken down to bicarbonates. The difference between them is that lactates are metabolized mainly in the liver while acetates are metabolized in all body cells. The latter is especially beneficial in liver insufficiency, lactic acidosis and microcirculation insufficiency leading to organ hypoperfusion.

ELIGIBILITY:
Inclusion Criteria:

* patients>18 years old, undergoing elective hepatobiliary surgery under general anesthesia and American Society of Anesthesiologists grade II.

Exclusion Criteria:

* 1-patient refusal. 2-psychiatric disorders. 3-pregnancy and lactation. 4-preexisting neurological dysfunction (history of cerebrovascular stroke CVS) 5-metastatic cancer. 6-Inflammatory bowel disease. 7-Diabetes mellitus. 8-Renal insufficiency (serum creatinine level more than 180 μmol/l). 9- unexpected intraoperative findings (inoperable). 10-accidental massive intraoperative hemorrhage.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2020-10-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
SGPT change pre- and postoperative | preoperative and in the first and second day postoperative
  effects of different fluid strategies in change of SGBT level pre- and postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Emad Zarief, assistant professor, Study Director — Assiut University